CLINICAL TRIAL: NCT06226948
Title: Using the Visualization for Lifestyle Change in Patients At Risk of Cardiovascular Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Maribor (Other)
Responsible Party: Principal Investigator, Adrijana Svensek, Principal Investigator, University Maribor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 05a/2I-2023
Record Dates: First submitted 2024-01-17; First posted 2024-01-26 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Cardiovascular Diseases; Coronary Artery Disease; Heart Diseases; Coronary Heart Disease; Visual Analytics; Continuous Glucose Monitoring; CGM; Lifestyle; Behaviour Change
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Artery Disease; Heart Diseases; Coronary Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Intervention group 1 (Experimental): Participants will use a continuous blood glucose monitoring and visualization of CVDs risk.
  Interventions: Device: CGM; Diagnostic Test: Visualization
- Intervention group 2 (Experimental): Participants will use a continuous blood glucose monitoring.
  Interventions: Device: CGM
- Intervention group 3 (Experimental): Participants will use a visualization of CVDs risk.
  Interventions: Diagnostic Test: Visualization
- Control group (No Intervention): No intervention.

INTERVENTIONS:
Device: CGM — Participants will wear CGM monitors for 10 days.
  Other Names: Intervention 1; Intervention 2
  Arms: Intervention group 1; Intervention group 2
Diagnostic Test: Visualization — Enriched visualization of SCORE2 CVD risk.
  Other Names: Intervention 1; Intervention 3
  Arms: Intervention group 1; Intervention group 3

SUMMARY:
In the framework of PhD research, the investigators will present a visualization of estimation of CVDs risk and the possibility of monitoring blood glucose levels in real-time. Based on the results, the investigators will assess the association of these with lifestyle change. The findings highlight the need for sufficiently reliable and high-quality evaluations of visualizations, technologies or applications used in the family medicine.

DETAILED DESCRIPTION:
The investigators reviewed the existing literature and found little research on the use of Continuous Glucose Monitoring (CGM) and visualization of SCORE2 prognostic model in healthy populations and how they can influence lifestyle change. The investigators will conduct a randomised control trial with 3 intervention groups and 1 control gropu. The investigators also found that primary care nurses are still using paper-based methods to calculate CVDs by using colour-coded charts. Therefore, the investigators will use the visual tool of the SCORE2 scale to identify possible increased participants motivation using visualization. The investigators will also confirm or refute lifestyle change by calculating biological age.

ELIGIBILITY:
Inclusion Criteria:

* individuals ages more than 40 years
* without serious disease progression
* at least one risk factor for CVDs

Exclusion Criteria:

* individuals younger than 40 years
* with serious disease progression
* without risk factor for CVDs

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-05-06 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
Assessment of change of lifestyle. | Change in Healthy Lifestyle and Personal Control Questionnaire score will be assessed at the enrolment of the participants followed by the examination in the period of up to 6 months after the enrolment.
  Change of lifestyle will be assessed using the Healthy Lifestyle and Personal Control Questionnaire from Darviri, et al., 2014. The goal of this questionnaire is to detect and quantify lifestyle patterns that reflect health empowerment and for assessing the efficacy of future health-promoting interventions to improve individuals' lifestyles and wellbeing.
  The assessment is based on a 4-point Likert scale (1 = never or rarely, 2 = sometimes, 3 = often and 4 = always). The final calculation of lifestyle is based on the sum of the dimensions. The dimensions can also be compared individually with each other at the final stage to determine which dimension has experienced the greatest change in lifestyle. The minimum possible score is 31, indicating no change in lifestyle, and the maximum possible score is 90, indicating the greatest change in lifestyle.
Assessment of person-centred care. | The Person-Centred Practice Inventory - Service User score will be assessed at the enrolment of the participants followed by the examination in the period of up to 6 months after the enrolment.
  The Person-Centred Practice Inventory - Service User consists of 20 items measuring participants agreement with statements related to perceptions of person-centred care and includes 5 constructs: working with participants beliefs and values, shared decision making, compassionate presence and holistic care.The score is based on a 5-point Likert scale. The lowest level of participants agreement is 20 and the highest level is 100.
Systematic Coronary Risk Evaluation 2 risk | Change in Systematic Coronary Risk Evaluation 2 score will be assessed at the enrolment of the participants followed by the examination in the period of up to 6 months after the enrolment.
  Systematic Coronary Risk Evaluation 2 is designed to calculate the risk of CVD according to the Systematic Coronary Risk Evaluation 2 prognostic model (ESC, 2022).The higher the percentage, the higher the risk.

SECONDARY OUTCOMES:
Assessment in Biological age | Change in Biological age will be assessed at the enrolment of the participants followed by the examination in the period of up to 3 and 6 months after the enrolment.
  Biological age tells us whether we are physiologically younger or older than our chronological age.The scale depends on each individual - it's individual. The closer the biological age result is to the chronological one, the better the result.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Health Sciences, Maribor, Slovenia

IPD SHARING:
Plan to Share IPD: No
The anonymity of all research participants will be guaranteed throughout the research. Only the researcher involved will have access to the anonymised data.

REFERENCES:
- [Background] Darviri C, Alexopoulos EC, Artemiadis AK, Tigani X, Kraniotou C, Darvyri P, Chrousos GP. The Healthy Lifestyle and Personal Control Questionnaire (HLPCQ): a novel tool for assessing self-empowerment through a constellation of daily activities. BMC Public Health. 2014 Sep 24;14:995. doi: 10.1186/1471-2458-14-995. PMID 25253039
- See also: European Society of Cardiology — https://www.escardio.org/Education/Practice-Tools/CVD-prevention-toolbox/SCORE-Risk-Charts